CLINICAL TRIAL: NCT01501773
Title: Phase II Intravenous Autologous Bone Marrow-derived Stem Cells Therapy for Patients With Acute Ischemic Stroke
Brief Title: Intravenous Autologous Bone Marrow-derived Stem Cells Therapy for Patients With Acute Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Manipal Acunova Ltd. (Network)
Collaborators: Ministry of Science and Technology, India (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INVEST
Record Dates: First submitted 2011-12-26; First posted 2011-12-29 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Acute Stroke
Keywords: Acute ischemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous bone marrow stem cell (Experimental)
  Interventions: Biological: Autologous bone marrow stem cell
- Control (No Intervention)

INTERVENTIONS:
Biological: Autologous bone marrow stem cell — Autologous bone marrow stem cell have bone marrow aspiration and receive 30-500 million bone marrow mononuclear cells intravenously on the day of randomization.
  Arms: Autologous bone marrow stem cell

SUMMARY:
A multi-centric initiative to study safety,feasibility and efficacy of using intravenous autologous bone marrow mononuclear cells(BMMC) in patients with acute ischemic stroke.This phase of study is visualised as phase 2 study and will aim to determine dose response gradient of stem cell therapy and to explore if there is favorable risk to benefit ratio for autologous stem cell therapy in patient with acute ischamic stroke.

DETAILED DESCRIPTION:
This phase of the study will have two arms developed through random allocation: one arm for intravenous autologous bone marrow derived stem cell/mononuclear cells(BMMC arm); and second control arm. Patients with acute ischaemic stroke between 7-30 days after onset with moderae severity in sable condition will be entered into the study after informed consent. Both arms will receive standard treatment but BMMC arm will,in addition,have bone marrow aspiration and receive autologous 30-500 million bone marrow mononuclear cells intravenously on the day of randomisation and all patients will be followed at DaY 7 ± days, Day 90(-7 days to +14 days), Day 180(-7 days to +28 days)and Day 365 (-7 days to + 28 days). A number of safety and efficacy variables will be measured. This phase 2 study will aim to determine dose response gradient of stem cell therapy and to explore if results have a favourable risk to benefit ratio to justify a phase 3 study. This will be the first human trial to determine and compare favourable and unfavourable effects of bone marrow mononuclear cells(mainly CD34) in acute ischamic stroke and also the first multi-centric study with potential to achieve a reasonable sample size in a relatively short time.

ELIGIBILITY:
Inclusion Criteria:

1. Sudden onset of focal neurologic deficit or impairment of consciousness.
2. CT or MRI scan of head showing no haematoma and relevant lesions within the MCA and ACA territory.
3. Age between 30 -70 years (after amendment 18 -70 years).
4. >7 to </=30 days passed since the onset of the qualifying event.
5. Glasgow Coma Scale score of >8 at the time of randomization, in aphasic Eye and Motor score of >6.
6. Modified Barthel Index score of 50 or less at the time of randomization.
7. NHISS score of 7 or more points and inability to walk unaided or raise upper limb by 90 degree.
8. Patient is stable. ( normal respiration, afebrile, BP less than mean arterial pressure of 125 mm of Hg, fasting blood sugar < 200 mg% and normal urea/electrolytes for at least 48 hours.)

Exclusion Criteria: -

1. Lacunar syndrome
2. Intubation
3. Posterior circulation stroke
4. Co morbidity likely to limit survival to less than 3 years eg. Hepatic or renal failure.
5. Inaccessibility for follow up.
6. Allergy to local anaesthetic.
7. Unwillingness to provide written informed consent.
8. Symptom of acute myocardial infarction or acute involvement of any other organ.
9. Pregnancy 10. HIV positive 11. Patient is a part of any other trial in last 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Barthel index score | six month post randomization
  The primary efficacy outcome is difference between the two groups in the modified Barthel index score at six month post randomization.

SECONDARY OUTCOMES:
NIHSS score and functional status | 3, 6 and 12 months post randomization
  1. NIHSS score at 6 months and one year post randomization.
  2. And degree of handicap as measured by Modified Ranking scale administered at 3, 6 and 12 months post randomization and functional status at 6 months and 12 months post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Kameshwar Prasad, MBBS, MD, Principal Investigator — All India Institute of Medical Sciences; Dr. Usha Kant Misra, MBBS, MD, DM, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences; Dr. R.S Sarkar, Principal Investigator — Armed Forces Medical College; Dr. Sudesh Kumar Prabhakar, MBBS, MD, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Dr. Sharat Joshi, MBBS,MD, DM, Principal Investigator — Army R & R Hospital
Locations (5):
- India (5):
  - Post Graduate Institute of Medical Education and Research, Chandīgarh, Haryana
  - Armed Forces Medical College, Pune, Maharashtra
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Army Hospital (R & R Hospital), New Delhi, National Capital Territory of Delhi
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh

REFERENCES:
- [Derived] Prasad K, Sharma A, Garg A, Mohanty S, Bhatnagar S, Johri S, Singh KK, Nair V, Sarkar RS, Gorthi SP, Hassan KM, Prabhakar S, Marwaha N, Khandelwal N, Misra UK, Kalita J, Nityanand S; InveST Study Group. Intravenous autologous bone marrow mononuclear stem cell therapy for ischemic stroke: a multicentric, randomized trial. Stroke. 2014 Dec;45(12):3618-24. doi: 10.1161/STROKEAHA.114.007028. Epub 2014 Nov 6. PMID 25378424
- [Derived] Prasad K, Mohanty S, Bhatia R, Srivastava MV, Garg A, Srivastava A, Goyal V, Tripathi M, Kumar A, Bal C, Vij A, Mishra NK. Autologous intravenous bone marrow mononuclear cell therapy for patients with subacute ischaemic stroke: a pilot study. Indian J Med Res. 2012 Aug;136(2):221-8. PMID 22960888